CLINICAL TRIAL: NCT02428751
Title: Rituximab, Cyclophosphamide, Vincristine, and Prednisone in Combination With Doxorubicin (R-CHOP) Versus in Combination With Pegylated-liposomal Doxorubicin (R-CDOP) as First-line Treatment for Elderly Patients With Diffuse Large-B-cell Lymphoma: a Randomised, Multicentre, Non-inferiority Study
Brief Title: R-CHOP Versus R-CDOP as First-line Treatment for Elderly Patients With Diffuse Large-B-cell Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenqi Jiang (Other)
Responsible Party: Sponsor-Investigator, Wenqi Jiang, Chief of Department of Internal Medicine, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 308-2015-005
Record Dates: First submitted 2015-04-17; First posted 2015-04-29 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: Lymphoma, Large B-Cell, Diffuse; liposomal doxorubicin; doxorubicin; event-free survival
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — liposomal doxorubicin; Doxorubicin; Rituximab; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- R-CHOP (Active Comparator): This group received R-CHOP regimen as the first-line chemotherapy. Rituximab, 375mg/m2, iv, d0; Cyclophophamide, 750mg/m2, iv, d1; Doxorubicin, 50mg/m2, iv, d1; Vincristine, 2mg/m2 (max 2mg), iv, d1; Prednisone, 100mg, po, d1-5. Repeat every 21 days for 6-8 cycles or until the criteria of terminating treatment was met.
  Interventions: Drug: Doxorubicin; Drug: Rituximab; Drug: Cyclophophamide; Drug: Vincristine; Drug: Prednisone
- R-CDOP (Experimental): This group received R-CDOP regimen as the first-line chemotherapy. Rituximab, 375mg/m2, iv, d0; Cyclophophamide, 750mg/m2, iv, d1; Pegylated liposomal doxorubicin, 30mg/m2, iv, d1; Vincristine, 2mg/m2 (max 2mg), iv, d1; Prednisone, 100mg, po, d1-5. Repeat every 21 days for 6-8 cycles or until the criteria of terminating treatment was met.
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Rituximab; Drug: Cyclophophamide; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin — 30 mg/m2, IV (in the vein) on day 1 of each 21 day cycle
  Arms: R-CDOP
Drug: Doxorubicin — 50 mg/m2, IV (in the vein) on day 1 of each 21 day cycle
  Arms: R-CHOP
Drug: Rituximab — 375 mg/m2, IV (in the vein) on day 0 of each 21 day cycle
Drug: Cyclophophamide — 750 mg/m2, IV (in the vein) on day 1 of each 21 day cycle
Drug: Vincristine — 1.4 mg/m2 (2mg in maxium), IV (in the vein) on day 1 of each 21 day cycle
Drug: Prednisone — 100mg/d, PO on day 1-5 of each 21 day cycle

SUMMARY:
The combination of rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP regimen) has been the first-line chemotherapy for elderly patients with diffuse large B-cell lymphoma (DLBCL). The treatment-related toxicities, especially the severe cardiac toxicities induced by anthracycline drugs (doxorubicin), have become a major concern among elderly patients. Pegylated liposomal doxorubicin is a formulation of doxorubicin with a prolonged circulation time and unique toxicity profile. Previous single arm studies of elderly patients with lymphoma used pegylated liposomal doxorubicin instead of traditional doxorubicin in combination with rituximab, cyclophosphamide, vincristine, and prednisone (the novel R-CDOP regimen), and demonstrated better safety profile, including less bone marrow suppression and less cardiac toxicities, while maintaining the efficacy. However, the efficacy and safety of these two regimens (R-CHOP and R-CDOP) have not been head-to-head compared in a randomized study. The aim of this study is to compare the efficacy and safety of R-CDOP (rituximab, cyclophosphamide, pegylated liposomal doxorubicin, vincristine, and prednisone) and R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone) in previously untreated elderly patients with DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of CD20-positive diffuse large B-cell lymphoma
* 60~80 years old
* Ann Arbor stage I~IV
* ECOG physical score of 0~2
* Have not received previous treatment to lymphoma, including chemotherapy, radiotherapy, or biotherapy
* Have at least one clinically measurable lesion: >= 2cm under physical examination, or >= 1.5cm under computed tomography (CT) or magnetic resonance (MR)
* Life expectancy of >= 3 months
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase and total bilirubin <= 2 × upper limit of normal (ULN)
* Glomerular filtration rate (MDRD method) >= 30ml/min
* No abnormalities in blood coagulative function
* Generally normal bone marrow function: while blood cell >= 3,000/μL, absolute neutrophil count >= 1,500/μL, hemoglobin >= 100g/L, platelet >= 75,000/μL
* No evidence of active hepatitis B or C virus, or human immunodeficiency virus infection
* Left ventricular ejection fraction (LVEF) >= 45% measured by two dimensional echocardiography or multi-gated acquisition (MUGA) scan
* Cardiac function of class I-II in New York Heart Association (NYHA) classification

Exclusion Criteria:

* Patients with indolent lymphoma
* Positive results for in situ hybridization for Epstein-Barr virus encoded RNA (EBER)
* Serum Epstein-Barr virus DNA >= 1,000 copies/ml
* Double-hit lymphoma confirmed by fluorescence in situ hybridization (FISH)
* Primary mediastinal B-cell lymphoma
* Involvement of central nervous system
* Bulky disease (>= 10cm)
* History of cardiac disease, including clinically significant ventricular tachycardia, atrial fibrillation, conduction block, myocardial infarction within 1 year, congestive heart failure, symptomatic coronary heart disease which needs medication
* Known allergic reaction to any component of the agents used in the chemotherapeutic regimens that are used in the study
* Previous exposure to anthracycline drugs, rituximab, or chemotherapy for lymphoma
* History of malignant carcinoma within 5 years (except carcinoma in situ of the skin and uterine cervix, and prostatic carcinoma)
* Currently enrolled in other clinical studies
* Other conditions that the investigators consider as inappropriate for enrolling into this study

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
event-free survival (EFS) | two year
  Defined as time from the date of randomization to the date of disease progression, death due to any cause, termination of treatment, or the most recent follow-up

SECONDARY OUTCOMES:
overall response rate (ORR) | at week 6, 12, 18, and 24 after randomization
  defined as the proportion of patients whose best overall response is either complete remission (CR) or partial remission (PR), which was evaluated in accordance with the International Working Group Recommendations for Response Criteria for non-Hodgkin's lymphoma
complete remission (CR) rate | at week 6, 12, 18, and 24 after randomization
  defined as the proportion of patients whose best overall response is complete remission, which was evaluated in accordance with the International Working Group Recommendations for Response Criteria for non-Hodgkin's lymphoma
overall survival (OS) | two year
  defined as time from the date of randomization to the date of death due to any cause or the most recent follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wen-qi Jiang, M.D., Principal Investigator — Sun Yat-sen University
Locations (7):
- China (7):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical Unversity, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Wujing Zongdui Hospital of Guangdong Province, Guangzhou, Guangdong

REFERENCES:
- [Result] Fisher RI, Gaynor ER, Dahlberg S, Oken MM, Grogan TM, Mize EM, Glick JH, Coltman CA Jr, Miller TP. Comparison of a standard regimen (CHOP) with three intensive chemotherapy regimens for advanced non-Hodgkin's lymphoma. N Engl J Med. 1993 Apr 8;328(14):1002-6. doi: 10.1056/NEJM199304083281404. PMID 7680764
- [Result] Feugier P, Van Hoof A, Sebban C, Solal-Celigny P, Bouabdallah R, Ferme C, Christian B, Lepage E, Tilly H, Morschhauser F, Gaulard P, Salles G, Bosly A, Gisselbrecht C, Reyes F, Coiffier B. Long-term results of the R-CHOP study in the treatment of elderly patients with diffuse large B-cell lymphoma: a study by the Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol. 2005 Jun 20;23(18):4117-26. doi: 10.1200/JCO.2005.09.131. Epub 2005 May 2. PMID 15867204
- [Result] Coiffier B, Thieblemont C, Van Den Neste E, Lepeu G, Plantier I, Castaigne S, Lefort S, Marit G, Macro M, Sebban C, Belhadj K, Bordessoule D, Ferme C, Tilly H. Long-term outcome of patients in the LNH-98.5 trial, the first randomized study comparing rituximab-CHOP to standard CHOP chemotherapy in DLBCL patients: a study by the Groupe d'Etudes des Lymphomes de l'Adulte. Blood. 2010 Sep 23;116(12):2040-5. doi: 10.1182/blood-2010-03-276246. Epub 2010 Jun 14. PMID 20548096
- [Result] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Result] Habermann TM, Weller EA, Morrison VA, Gascoyne RD, Cassileth PA, Cohn JB, Dakhil SR, Woda B, Fisher RI, Peterson BA, Horning SJ. Rituximab-CHOP versus CHOP alone or with maintenance rituximab in older patients with diffuse large B-cell lymphoma. J Clin Oncol. 2006 Jul 1;24(19):3121-7. doi: 10.1200/JCO.2005.05.1003. Epub 2006 Jun 5. PMID 16754935
- [Result] Limat S, Daguindau E, Cahn JY, Nerich V, Brion A, Perrin S, Woronoff-Lemsi MC, Deconinck E. Incidence and risk-factors of CHOP/R-CHOP-related cardiotoxicity in patients with aggressive non-Hodgkin's lymphoma. J Clin Pharm Ther. 2014 Apr;39(2):168-74. doi: 10.1111/jcpt.12124. Epub 2014 Jan 3. PMID 24384030
- [Result] Gogas H, Papadimitriou C, Kalofonos HP, Bafaloukos D, Fountzilas G, Tsavdaridis D, Anagnostopoulos A, Onyenadum A, Papakostas P, Economopoulos T, Christodoulou C, Kosmidis P, Markopoulos C. Neoadjuvant chemotherapy with a combination of pegylated liposomal doxorubicin (Caelyx) and paclitaxel in locally advanced breast cancer: a phase II study by the Hellenic Cooperative Oncology Group. Ann Oncol. 2002 Nov;13(11):1737-42. doi: 10.1093/annonc/mdf284. PMID 12419745
- [Result] Tulpule A, Espina BM, Berman N, Buchanan LH, Smith DL, Sherrod A, Dharmapala D, Gee C, Boswell WD, Nathwani BN, Welles L, Levine AM. Phase I/II trial of nonpegylated liposomal doxorubicin, cyclophosphamide, vincristine, and prednisone in the treatment of newly diagnosed aggressive non-Hodgkin's lymphoma. Clin Lymphoma Myeloma. 2006 Jul;7(1):59-64. doi: 10.3816/CLM.2006.n.040. PMID 16879771
- [Result] O'Brien ME, Wigler N, Inbar M, Rosso R, Grischke E, Santoro A, Catane R, Kieback DG, Tomczak P, Ackland SP, Orlandi F, Mellars L, Alland L, Tendler C; CAELYX Breast Cancer Study Group. Reduced cardiotoxicity and comparable efficacy in a phase III trial of pegylated liposomal doxorubicin HCl (CAELYX/Doxil) versus conventional doxorubicin for first-line treatment of metastatic breast cancer. Ann Oncol. 2004 Mar;15(3):440-9. doi: 10.1093/annonc/mdh097. PMID 14998846
- [Result] Luminari S, Montanini A, Caballero D, Bologna S, Notter M, Dyer MJS, Chiappella A, Briones J, Petrini M, Barbato A, Kayitalire L, Federico M. Nonpegylated liposomal doxorubicin (MyocetTM) combination (R-COMP) chemotherapy in elderly patients with diffuse large B-cell lymphoma (DLBCL): results from the phase II EUR018 trial. Ann Oncol. 2010 Jul;21(7):1492-1499. doi: 10.1093/annonc/mdp544. Epub 2009 Dec 11. PMID 20007997
- [Result] Corazzelli G, Frigeri F, Arcamone M, Lucania A, Rosariavilla M, Morelli E, Amore A, Capobianco G, Caronna A, Becchimanzi C, Volzone F, Marcacci G, Russo F, De Filippi R, Mastrullo L, Pinto A. Biweekly rituximab, cyclophosphamide, vincristine, non-pegylated liposome-encapsulated doxorubicin and prednisone (R-COMP-14) in elderly patients with poor-risk diffuse large B-cell lymphoma and moderate to high 'life threat' impact cardiopathy. Br J Haematol. 2011 Sep;154(5):579-89. doi: 10.1111/j.1365-2141.2011.08786.x. Epub 2011 Jun 28. PMID 21707585
- [Result] Zaja F, Tomadini V, Zaccaria A, Lenoci M, Battista M, Molinari AL, Fabbri A, Battista R, Cabras MG, Gallamini A, Fanin R. CHOP-rituximab with pegylated liposomal doxorubicin for the treatment of elderly patients with diffuse large B-cell lymphoma. Leuk Lymphoma. 2006 Oct;47(10):2174-80. doi: 10.1080/10428190600799946. PMID 17071492
- [Result] Rigacci L, Mappa S, Nassi L, Alterini R, Carrai V, Bernardi F, Bosi A. Liposome-encapsulated doxorubicin in combination with cyclophosphamide, vincristine, prednisone and rituximab in patients with lymphoma and concurrent cardiac diseases or pre-treated with anthracyclines. Hematol Oncol. 2007 Dec;25(4):198-203. doi: 10.1002/hon.827. PMID 17654614
- [Result] Visani G, Guiducci B, D'Adamo F, Mele A, Nicolini G, Leopardi G, Sparaventi G, Barulli S, Malerba L, Isidori A, Malagola M, Piccaluga PP. Cyclophosphamide, pegylated liposomal doxorubicin, vincristine and prednisone (CDOP) plus rituximab is effective and well tolerated in poor performance status elderly patients with non-Hodgkin's lymphoma. Leuk Lymphoma. 2005 Mar;46(3):477-9. doi: 10.1080/10428190400013688. No abstract available. PMID 15621843
- [Result] Heintel D, Skrabs C, Hauswirth A, Eigenberger K, Einberger C, Raderer M, Sperr WR, Knobl P, Mullauer L, Uffmann M, Dieckmann K, Gaiger A, Jager U. Nonpegylated liposomal doxorubicin is highly active in patients with B and T/NK cell lymphomas with cardiac comorbidity or higher age. Ann Hematol. 2010 Feb;89(2):163-9. doi: 10.1007/s00277-009-0796-5. Epub 2009 Jul 28. PMID 19636553
- [Result] Gimeno E, Sanchez-Gonzalez B, Alvarez-Larran A, Pedro C, Abella E, Comin J, Saumell S, Garcia-Pallarols F, Gomez M, Besses C, Salar A. Intermediate dose of nonpegylated liposomal doxorubicin combination (R-CMyOP) as first line chemotherapy for frail elderly patients with aggressive lymphoma. Leuk Res. 2011 Mar;35(3):358-62. doi: 10.1016/j.leukres.2010.07.024. Epub 2010 Aug 12. PMID 20708263